CLINICAL TRIAL: NCT00333567
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Compare Efficacy of a Single Dose of Lumiracoxib 400 mg Given Pre-Emptively Versus Post-Operatively, in Reducing Pain Associated With Ambulatory Arthroscopic Knee Surgery
Brief Title: Efficacy and Safety of Lumiracoxib 400 mg in Arthroscopic Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2427
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Pain
Keywords: arthroscopic knee surgery; cyclooxygenase-2 inhibitors; lumiracoxib; COX189; Ambulatory arthroscopic knee surgery
MeSH Terms: conditions — Pain | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study is designed to investigate the efficacy and safety of a single daily dose of 400 mg lumiracoxib given pre-emptively versus post-operatively in terms of efficacy in reducing pain associated with ambulatory arthroscopic knee surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients who need scheduled minor ambulatory arthroscopic knee surgery.

Exclusion Criteria:

* Patients with any surgical or medical conditions which could place the patient at higher risk from his/her participation in the study, or are likely to prevent the patient from complying with the requirements of the study or completing the trial period.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2006-08

PRIMARY OUTCOMES:
Pain Intensity (PI) in the target knee after movement at the 2 h time-point

SECONDARY OUTCOMES:
PI at 1, 2, 3, 4 and 24 h time-points while at rest
PI at 1, 3, 4 and 24 h time-points after movement
Time to first rescue medication intake
Patient's global evaluation of response to study medication
Safety and tolerability profile

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Director — Novartis
Locations (1):
- Novartis, Nuremberg, Germany